CLINICAL TRIAL: NCT04670731
Title: Study of Ventricular Remodelling and Metabolomics in Pediatric Cardiomyopathies (PROGRESS-OMICS)
Brief Title: Ventricular Remodelling and Metabolomics in Pediatric Cardiomyopathies (PROGRESS-OMICS)
Acronym: PRO-OMICS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Collaborators: Parent Project, Italy (Other); Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2259
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-11

CONDITIONS: Cardiomyopathies; Pediatric ALL
MeSH Terms: conditions — Cardiomyopathies; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples; endomyocardial specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The pathogenesis of cardiomyopathies is complex and a simple approach cannot describe the whole picture. Different etiologies are reported in pediatric age and heart failure onset can lead to poor prognosis in term of need of heart transplantation and ventricular assist device implantation. Based on hypothesis that heart failure development is related to heart inability to meet metabolic demands of the body, our study will focus to evaluate cardiac metabolism as one of the most critical factors and the accompanying changes of metabolic and echocardiographic profiles at different stages of heart failure. The heart is a unique organ working continuously as a pump supplying blood to the body. To meet this requirement, the myocardium utilizes fatty acids to generate 70-90% of the adenosine triphospate, with the rest being produced by oxidation of glucose, lactate, ketone bodies, aminoacids. Utilization of fatty acids is reduced in the failing heart and there is a metabolic shift to generation of adenosine triphospate from glucose. In patients with advanced cardiomyopathies, the heart is unable to utilize either metabolite and thus "runs out of fuel". It is reported that the adenosine triphospate level is approximately 30% lower in failing human hearts compared with non-failing hearts. In addition to this premise about the metabolic profile of the failing heart, recent advances in the field of metabolomics have indicated that several metabolites and/or metabolic pathways have a role in heart failure. Metabolism of lipids, glycolysis, fructolysis, aminoacids, and ketone oxidation have been found to be altered in non-ischemic cardiomyopathy in adult population. Also in adult heart failure patients some metabolic profiles resulted pronounced perturbated. Taking advantage of the high throughput, metabolomics is a platform for identifying metabolic signatures in children at each stages of heart failure (from pre clinical heart failure to end stage forms). We also will determine whether metabolomic analysis provides sensitive evaluation of heart failure in terms of remodelling at different stages and in disease regression after therapeutic interventions. Study desing is conceived in two parts. The first part is retrospective and we will analyze all echocardiograms in all children affected by cardiomyopathies. The second part is a cross sectional study in which will evaluate untargeted metabolomics in children at any stage of heart failure (A,B, C, D) and in control group. We will evaluate the clinical applicability and significance of plasma metabolomic analysis in the diagnosis and prognosis of heart failure in pediatric ages.

ELIGIBILITY:
Patients with Cardiomyopathies

Inclusion Criteria:

* Dilated Cardiomyopathy, defined as left ventricular dilation > 2SD
* A-D stages of Heart Failure, according to ACC/AHA definition
* < 18 years

Exclusion Criteria:

* Restrictive cardiomyopathy
* Hypertrophic cardiomyopathy
* Congenital Heart Diasease
* Valvular Heart Disease, as primary cause of heart failure
* > 18 years

Control Group

Inclusion Criteria:

* Children without familial disease and/ or abnormalities of ECG and echocardiographic, NT pro BNP ≥ 103 pg/mL, TnT ≥ 14

Exclusion Criteria:

* Children with familial disease and/or any abnormalities of ECG and echocardiographic abnormalities, NT pro BNP ≥ 103 pg/mL, TnT ≥ 14

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population will include all children (< 18 years) presenting with dilated cardiomyopathy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Identification of untargeted metabolomic profiles | 1 year
  Identification of metabolomic profiles in children with heart failure according to different stages od heart failure (A, predisposing condition; B- asymptomatic stage; C- symptomatic; D: end stage) and control group

SECONDARY OUTCOMES:
metabolomic profile and ventricular remodelling | 1 year
  correlation between metabolomic profiles and echocardiographic characteristic, such as left ventricular mass, left ventricular dilatation, mass/volume ratio) according to different stages of heart failure (A, predisposing condition; B- asymptomatic stage; C- symptomatic; D: end stage)
metabolomic profile and ventricular remodelling | 1 year
  correlation between metabolomic profiles and ECG characteristics, such as duration of PR, QRS, T wave change, according to different stages of heart failure (A, predisposing condition; B- asymptomatic stage; C- symptomatic; D: end stage)
identification of potential diagnostic of metabolomic profile | 1 year
  correlation between metabolomic profiles and clinical outcome, such as clinical stage, progression of remolling, death, heart transplantion, acute hospitalization for heart failure, VAD implantation, heart transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Rachele Adorisio, MD, Study Chair — Bambino Gesù Hospital and Research Institute, Rome, Italy; Rachele Adorisio, MD, Principal Investigator — Bambino Gesù Hospital and Research Institute, Rome, Italy
Locations (1):
- Bambino Gesù Hospital and Research Institute, Rome, Italy